CLINICAL TRIAL: NCT00359151
Title: Multicenter, Double Blind, Randomized, Placebo Controlled Trial Of The Efficacy And Safety Of Usual Care Plus Celecoxib Compared To Placebo For Peri-Operative And Rehabilitation Pain Control And Return To Function In Osteoarthritis Patients Undergoing Total Knee Arthroplasty
Brief Title: Celebrex Total Knee Arthroplasty Study
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: This study was terminated early due to slow enrollment.
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A3191225
Record Dates: First submitted 2006-07-28; First posted 2006-08-01 (Estimated); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Osteoarthritis; Pain
Keywords: Perioperative care of total arthroplasty assessing opioid consumption
MeSH Terms: conditions — Osteoarthritis; Pain | interventions — Celecoxib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Celecoxib (Experimental): Celecoxib
  Interventions: Drug: Celecoxib
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Celecoxib — 7 days pre-surgery (excluding day of surgery): 1 celecoxib 200 mg capsule or matching placebo QD; Day of surgery: 2 celecoxib 200 mg capsules or matching placebo within 2 hours prior to surgery, and 1 celecoxib 200 mg capsule or matching placebo following surgery; Post-surgery: starting the day after surgery, 1 celecoxib 200 mg capsule or matching placebo BID for the duration of the study.
  Arms: Celecoxib
Drug: Placebo — Placebo once daily (QD) for 7 days pre-surgery (excluding the day of surgery); Placebo within 2 hours prior to surgery; and post surgery on the same day of the surgery; Placebo twice daily (BID) following the day of surgery and for the duration of the study.
  Arms: Placebo

SUMMARY:
This study will investigate the benefits of administering celecoxib (Celebrex), a selective cyclooxygenase -2 (COX-2) inhibitor, in treating osteoarthritis (OA) subjects undergoing elective unilateral primary total knee arthroplasty (TKA) from the pre-operative phase to the management of post total knee replacement pain, and through the 6 weeks of physical therapy and rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* The subject is a male or female 18 years or older with osteoarthritis of the knee scheduled to undergo elective unilateral primary total knee arthroplasty because of OA, performed under a standardized regimen of anesthesia and procedure.

Exclusion Criteria:

* Subject has a history of inflammatory arthritis (e.g. rheumatoid arthritis, ankylosing spondylitis) other than osteoarthritis.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2006-11; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
To assess the effects of celecoxib on the cumulative amount of opioid administered to OA subjects undergoing unilateral total knee arthroplasty. | 19 July 2007

SECONDARY OUTCOMES:
To assess the effects of celecoxib on pain and function during the peri-operative period and the post-operative rehabilitation phase. | 19 July 2007
To assess the safety and tolerability of celecoxib in this study population. | 19 July 2007

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (6):
- United States (6):
  - Pfizer Investigational Site, Aurora, Colorado
  - Pfizer Investigational Site, Englewood, Colorado
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
  - Pfizer Investigational Site, Bellaire, Texas
  - Pfizer Investigational Site, Houston, Texas

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3191225&StudyName=Celebrex%20Total%20Knee%20Arthroplasty%20Study